CLINICAL TRIAL: NCT05116761
Title: Bone Marrow Mesenchymal Stem Cell Derived Extracellular Vesicles Infusion Treatment for Post-Acute and Chronic Post-COVID-19 Syndrome: A Phase I/II Clinical Trial
Brief Title: ExoFlo™ Infusion for Post-Acute COVID-19 and Chronic Post-COVID-19 Syndrome
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study no longer part of development plan.
Sponsor: Direct Biologics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DB-EF-POSTCOVID-0002
Record Dates: First submitted 2021-11-09; First posted 2021-11-11 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Covid19; Postviral Syndrome; Dyspnea
MeSH Terms: conditions — COVID-19; Dyspnea | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm 1 (Placebo Comparator): Normal Saline 100 mL
  Interventions: Other: Saline
- Treatment Arm 2 (Experimental): Normal saline 85 mL and ExoFlo 15 mL, which is 10.5 x 10^8 EV
  Interventions: Biological: Bone Marrow Mesenchymal Stem Cell Derived Extracellular Vesicles

INTERVENTIONS:
Biological: Bone Marrow Mesenchymal Stem Cell Derived Extracellular Vesicles — Intravenous administration of Bone Marrow Mesenchymal Stem Cell Derived Extracellular Vesicles
  Arms: Treatment Arm 2
Other: Saline — Placebo Saline
  Arms: Treatment Arm 1

SUMMARY:
This is a Phase I/II trial to evaluate the safety and efficacy of intravenous (IV) administration of bone marrow mesenchymal stem cell derived extracellular vesicles (EV), ExoFlo, as treatment for Post-Acute COVID-19 and Chronic Post-COVID-19 syndrome.

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of intravenous (IV) administration of bone marrow mesenchymal stem cell derived extracellular vesicles (EV), ExoFlo, as treatment for Post-Acute COVID-19 and Chronic Post-COVID-19 syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form (either by the individual or by the individual's healthcare proxy).
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female aged 18-85.
4. Discharged from recent hospitalization for severe COVID-19 disease requiring supplemental oxygen but not requiring mechanical ventilation or ECMO or dialysis.
5. Must be between 4 to 20 weeks since onset of acute COVID-19 symptoms onset.
6. No return to baseline health or hiatus between acute COVID-19 and onset of post-acute COVID-19 or chronic post-COVID-19 syndrome.
7. Current SARS-CoV-2 RT PCR must be negative prior to enrollment.
8. At least 2 or more persistent symptoms frequently reported for post-acute COVID-19 or chronic post-COVID-19 syndrome such as fatigue, cough, headache, body aches, fever, chills, loss of taste, loss of smell, diarrhea, congestion, dyspnea, sore throat, chest pain, abdominal pain, confusion, or vomiting must be moderate in severity based on modified CDC Symptoms Questionnaire (See Section 11.1 for severity scoring system).
9. Medical Resource Council Dyspnea Score of < 3 out of 5.
10. Baseline EQ-5D-5L must be higher than 21211. (Of note: EQ-5D-5L has 5 dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each dimension is scored from 1 (full) to 5 (worst), such that a score of 11111 is reflective of full quality-of-life and a score of 55555 is reflective of worst quality-of-life.)
11. Baseline 6-Minute Walk Test (6-MWT) is 500 meters or less.
12. Supplemental oxygen should be ≤5 L O2/min.
13. If the candidate is either male or female of reproductive potential, he or she must agree to use of double barrier method of highly effective birth control contraception such as condoms with oral contraceptive pill or choose to remain abstinent if already practicing abstinence during the screening period. The duration of required usage of double barrier method OR maintenance of abstinence must include the time from the beginning of the screening period until 90 days following the last dose of the study treatment.

Exclusion Criteria:

1. Vulnerable populations such as pregnant patients, children, individuals with severe physical or mental disabilities who cannot provide meaningful consent.
2. Active malignancy requiring treatment within the last five years.
3. Major physical trauma in the last 3 months, including motor vehicle accidents, assaults, mechanical falls with sequelae of significant bleeding or craniofacial bruising, and surgeries.
4. Patients with persistent symptoms due to any of the following chronic comorbidities such as active tuberculosis or cystic fibrosis, chronic respiratory disease including chronic obstructive pulmonary disease or pulmonary fibrosis requiring baseline home oxygen > 5 L O2/min, history of unstable angina or a heart attack during the last 12 months, pulmonary hypertension, hepatic impairment, chronic kidney disease, uncontrolled diabetes, substance abuse, severe osteoarthritis, HIV, migraine disorder, fibromyalgia, dementia, connective tissue disorders, and endocrine disorders.
5. Depression as screened by positive Patient Health Questionnaire (PHQ2) and confirmed as moderate or higher severity on PHQ9 (See Appendix 11.5). Of note, subjects found to have moderate or higher on PHQ-9 will be referred for appropriate outpatient psychiatric evaluation and intervention for their depression.
6. Vital sign abnormalities: temperature ≥ 38 °C, temperature < 35 °C; systolic blood pressure (SBP) < 90 mmHg, SBP ≥ 170 mmHg; diastolic blood pressure (DBP) < 50 mmHg, DBP ≥ 100 mmHg; heart rate (HR) < 50 beats per minute (BPM), HR ≥ 120 BPM.
7. Lab abnormalities: WBC ≥ 12,000 /μL, Creatinine ≥ 1.5 mg/dL, AST ≥ 100 IU/l, and/or ALT ≥ 100 IU/I
8. Patients who require rolling walker or wheelchair or higher level of assistance for ambulation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Increased distance on Six Minute Walk Test (6MWT) | 61 Days
  Meters walked in a self-paced test in which the subject is instructed to walk as fast as possible during 6 minutes.
Incidence of Serious Adverse Events (SAEs) | 61 Days
  Rate of SAEs observed over the duration of the study.

SECONDARY OUTCOMES:
EuroQol-5D (EQ-5D) | 61 days
  Five dimensions include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression
Medical Research Council (MRC) Dyspnea Scale | 61 Days
  Degree of breathlessness related to activity, graded 1-5.

OTHER OUTCOMES:
C-Reactive Protein (CRP), D-dimer, Atrial Natriuretic Peptides (ANP) | 61 Days
  Acute phase reactants

CONTACTS AND LOCATIONS:
Overall Officials: Bill Arana, Study Director — Direct Biologics, LLC